CLINICAL TRIAL: NCT01861158
Title: Online Parent Training for Children With Behavior Disorders: Phase II
Brief Title: Online Parent Training for Children With Behavior Disorders
Acronym: PW2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Family Works Incorporated (Other)
Collaborators: Oregon Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 2R44DA026658-02A1 (NIH)
Record Dates: First submitted 2013-05-20; First posted 2013-05-23 (Estimated); Last update posted 2017-02-14 (Actual); Status verified 2017-02

CONDITIONS: Parenting; Delinquency
Keywords: Parenting; Adolescence; Delinquency; Online intervention; Juvenile Justice

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Parenting Wisely (Experimental): Immediate access to the online Parenting Wisely program
  Interventions: Behavioral: Parenting Wisely
- Parenting Wisely + Community Forum (Active Comparator): Immediate access to the online Parenting Wisely program, as well as access to a community form where parents can receive social support from other online users of the program and a moderator
  Interventions: Behavioral: Parenting Wisely
- Delayed Parenting Wisely (No Intervention): Delayed (6-month) access to the Parenting Wisely program. Parents will receive access to PW after the final, 6-month, follow-up assessment.

INTERVENTIONS:
Behavioral: Parenting Wisely — Computer-based, online, interactive parenting intervention
  Other Names: PW
  Arms: Parenting Wisely; Parenting Wisely + Community Forum

SUMMARY:
This study evaluates Parenting Wisely (PW), an interactive, computer-based, online parenting program, through a formal randomized trial conducted in collaboration with the juvenile justice system (JJS), the primary market for such a program. Parents of 450 delinquent receiving JJS services as usual (SAU) will be randomly assigned to: PW plus a social networking online discussion forum, PW alone, or SAU. The investigators will also determine the potential marketability of the PW intervention to JJS programs based on the effects of PW on parent report and direct observation measures of parenting behaviors, adolescent behaviors, and family functioning, as well as measures of recidivism and cost savings. User satisfaction, program comprehension, receptivity, and parent self-efficacy will also be assessed. The investigators hypothesize that the two PW interventions (PW only and PW + Social Network) will produce greater reductions in disruptive behavior problems from baseline to 3- and 6-month assessments compared to SAU.

DETAILED DESCRIPTION:
Research has shown that parent-targeted interventions are effective in ameliorating adolescent conduct disorders, substance abuse, HIV-risk, and related adolescent problem behaviors. The meteoric rise of Internet use and recent advance in multimedia technology and software combine to create new opportunities for disseminating evidence-based practices. Parenting Wisely (PW; Gordon, 2000) is a computer-based intervention designed to prevent and treat child disruptive behavior problems. This evidence-based approach fits easily into existing juvenile justice, health, education, and mental health service delivery systems, bypassing many of the current barriers to care. The investigators' Phase I study focused on revising and enhancing PW with more culturally relevant content and imagery to broaden its appeal to ethnically diverse populations. The findings revealed substantial improvements on virtually all measures of parenting and child behavior and outcomes at 6 months were highly significant and clinically meaningful. This Phase II study is designed to broaden the appeal and potential reach of PW through a formal randomized trial conducted in collaboration with the juvenile justice system (JJS), the primary market for such a program. Parents of 450 delinquent receiving JJS services as usual (SAU) will be randomly assigned to: PW plus a social networking online discussion forum, PW alone, or SAU. PW is the first online skill-building parent training program to examine effectiveness across different ethnic cultural groups and offers a brief, low cost, accessible approach that could be easily and quickly implemented and sustained in JJS settings. As such, the potential impact for marketing PW and reducing child behavior problems is considerable. Phase II activities will include the development of a moderated online forum to increase parental social support and skill acquisition. The investigators will also determine the potential marketability of the PW intervention to JJS programs based on the effects of PW on parent report and direct observation measures of parenting behaviors, adolescent behaviors, and family functioning, as well as measures of recidivism and cost savings. User satisfaction, program comprehension, receptivity, and parent self-efficacy will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Parent of a 12-17 year old adolescent who has been referred to the juvenile justice system for a legal offense (at least one police-generated report)
* Adolescent has been referred by a participating county in Oregon or Nevada
* Parent and adolescent live together at least 40% of the time

Exclusion Criteria:

* Parent has already enrolled or completed the study for another adolescent
* Read and speak a language other than English or Spanish

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 306 (Actual)
Dates: Start 2012-09; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Parenting skills and knowledge | Change from baseline to 6-month follow-up
  Online questionnaire measures (Family Assessment Device, Parenting Scale, Parenting Knowledge Test, Parent Sense of Competence, Social Support for Parenting)
Child behavioral changes | Change from baseline to 6-month follow-up
  Online questionnaires (Eyberg Child Behavior Inventory, Strengths & Difficulties Questionnaire).
  Juvenile justice recidivism data for youth of the enrolled parents (e.g., new charges)

SECONDARY OUTCOMES:
Satisfaction with the Parenting Wisely program | 3 months following baseline
  Online questionnaires about program usability and user satisfaction: System Usability Scale and questions specific to parents' experiences with PW.

CONTACTS AND LOCATIONS:
Overall Officials: Don Gordon, Ph.D., Principal Investigator — Family Works Inc.
Locations (1):
- Oregon Research Institute, Portland, Oregon, United States